CLINICAL TRIAL: NCT03790982
Title: A Randomized, Double Blind, Placebo Controlled, Parallel-Group 52-week Multicenter Phase II Study to Investigate the Safety, Efficacy and Pharmacokinetics of AD-35 Tablet in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Evaluate the Safety and Efficacy of AD-35 Tablet in Subjects With Mild to Moderate Alzheimer's Disease
Acronym: WAY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-35-II-01
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer's Disease
Keywords: AD-35 tablet; Alzheimer's Disease; Phase II study
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Multiple Groups, Multiple Centers
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo of AD-35 60mg /AD-35 30mg (Placebo Comparator): Placebo of AD-35 60 mg Placebo of AD-35 30mg x two tablets, once daily in the first 26 weeks (oral), then AD-35 30mg +Placebo of AD-35 30mg, once daily in the second 26 weeks (oral)
  Interventions: Drug: Placebo of AD-35 60mg /AD-35 30mg
- Placebo of AD-35 60mg /AD-35 60mg (Placebo Comparator): Placebo of AD-35 60 mg Placebo of AD-35 30mg x two tablets, once daily in the first 26 weeks (oral), then AD-35 30mg x two tablets, once daily in the second 26 weeks (oral)
  Interventions: Drug: Placebo of AD-35 60mg /AD-35 60mg
- AD-35 30 mg+Placebo of AD-35 30 mg (Experimental): AD-35 30 mg + Placebo of AD-35 30 mg AD-35 30 mg + Placebo of AD-35 30 mg, once daily for 52 weeks (oral)
  Interventions: Drug: AD-35 30 mg + Placebo of AD-35 30 mg
- AD-35 60 mg (Experimental): AD-35 60 mg AD-35 30 mg× two tablets, once daily for 52 weeks (oral)
  Interventions: Drug: AD-35 60 mg

INTERVENTIONS:
Drug: Placebo of AD-35 60mg /AD-35 30mg — Placebo 60mg, oral, 1st 26 weeks; AD-35 30mg +Placebo of AD-35 30mg oral 2nd 26 weeks.
  Other Names: Placebo of AD-35
  Arms: Placebo of AD-35 60mg /AD-35 30mg
Drug: Placebo of AD-35 60mg /AD-35 60mg — Placebo 60mg, oral, 1st 26 weeks; AD-35 60mg oral, 2nd 26 weeks.
  Other Names: Placebo 60mg
  Arms: Placebo of AD-35 60mg /AD-35 60mg
Drug: AD-35 30 mg + Placebo of AD-35 30 mg — AD-35 30 mg + Placebo of AD-35 30 mg AD-35 30 mg + Placebo of AD-35 30 mg, Oral, 52 weeks.
  Other Names: AD-35
  Arms: AD-35 30 mg+Placebo of AD-35 30 mg
Drug: AD-35 60 mg — AD-35 60 mg AD-35 30 mg x two tablets, oral, 52 weeks.
  Other Names: AD-35
  Arms: AD-35 60 mg

SUMMARY:
Brief summary: This is a phase II study to investigate the safety, preliminary efficacy and pharmacokinetics of AD-35 tablet in patients with mild to moderate Alzheimer's Disease. This study is to be run in China involving 21 sites. It will enroll approximately 480 patients to ensure 240 randomized with mild to moderate Alzheimer's Disease. The treatment period is 52 weeks and total study duration per patient is approximately 57 weeks.

DETAILED DESCRIPTION:
In this multicenter, randomized, double blind, parallel-group, placebo controlled phase II study, 240 patients with mild to moderate Alzheimer's Disease are planned to be enrolled and randomly assigned 1:1:1 to receive placebo, or different doses of AD-35 tablet (30 or 60 mg). After the first 26 weeks, subjects on active study drug will remain on the current doses, and subjects assigned to placebo will be randomized to receive 30 mg and 60 mg AD-35 tablet in a 1:1 ratio, respectively, for the second 26 weeks. This study will evaluate the safety, preliminary efficacy and pharmacokinetics of AD-35 tablets in patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 50-75 years of age.
* Formal education of five or more years.
* Diagnosed of probable AD in accordance with the NINCDS/ADRDA criteria (2011).
* Mild or moderate AD subjects: MMSE Score of 15-26 and CDR Score ≥ 0.5 (CDR memory score ≥ 0.5).
* Subjects must have a brain magnetic resonance imaging (MRI) scan that is consistent with a clinical diagnosis of probable AD. Brain atrophy and medial temporal lobe atrophy visual assessment scale MTA grading >2 points. Mild white matter degeneration may occur, but Fazekas less than or equal to 2 points and supratentorial lacunar infarction lesions less than or equal to 3 points.
* The total score of modified Hachinski ischemia scale (MHIS) ≤ 4.
* Hamilton depression scale (HAMD) has a total score ≤ 17.

Exclusion Criteria:

* Visual, hearing and verbal communication of subjects cannot meet the needs of cognitive function evaluation.
* Inability to tolerate MRI procedures or contraindication to MRI, (such as implanted in the body, MRI incompatible pacemakers, implantable cardioverter defibrillators, cochlear implants, aneurysm clips, implanted injection pump, implanted nerve stimulator, metallic splinters in the eye, other magnetic, electrical and other metal implants) [note], or any other situation, in the judgment of the Investigator, is not suitable for magnetic resonance imaging (MRI).
* The investigators believe that other severe or unstable conditions may interfere with the cognitive evaluation in clinical trials.
* Dementia caused by other reasons: vascular dementia, central nervous system infection, endocrine system diseases (such as thyroid disease, parathyroid gland disease) and other reasons.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) 11 scores | Week 26
  Changes in the total of ADAS-Cog11 scores of treatment compared with baseline. The score ranged from 0 to 75, and the higher the score, the greater the cognitive impairment
Changes in Alzheimer's Disease Cooperative Study-clinical global impression of change (ADCS-CGIC ) scores | Week 26
  Changes in ADCS-CGIC scores of treatment compared with baseline. The overall condition of the disease change is assessed (improved or deteriorated) by the doctor and the patient, and the 8-point scoring method (0-7 points) was adopted.

SECONDARY OUTCOMES:
Changes in ADAS-Cog11 scores | Week 6, week 13, week 39, week52
  Changes in ADCS-CGIC scores of treatment compared with baseline

OTHER OUTCOMES:
Changes in ADCS-CGIC scores | Week 6, week 13, week 39, week52
  Changes in ADCS-CGIC scores of treatment compared with baseline
Changes in Mini-mental state examination (MMSE) scores | Week 6, week 13, week 26, week 39, week52
  Changes in MMSE scores of treatment compared with baseline. Each item has a correct score of 1 and an error score of 0.The total score ranges from 0 to 30, and the normal and abnormal boundary values are related to education degree. The lower the boundary value was the cognitive impairment, and the above was normal.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, PhD, Principal Investigator — Xuanwu hospital, capital medical university, Beijing, China
Locations (1):
- The Department of Neurosurgery, Beijing, Beijing Municipality, China